CLINICAL TRIAL: NCT05715138
Title: A Randomized Controlled Trial Comparing PAllidal and SubThalamic Deep Brain Stimulation for Cervical Dystonia（the PASTS-CD Study）
Brief Title: Comparison of Pallidal With Subthalamic Deep Brain Stimulation for Cervical Dystonia
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Zhiqi Mao, Professor, Chinese PLA General Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ChinaPLAGH_LB
Record Dates: First submitted 2023-01-10; First posted 2023-02-06 (Actual); Last update posted 2023-07-21 (Actual); Status verified 2023-07

CONDITIONS: Cervical Dystonia
Keywords: globus pallidus internus; subthalamic nucleus; deep brain stimulation
MeSH Terms: conditions — Torticollis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GPi-DBS (Experimental): The DBS electrodes are implanted into posteroventral GPi bilaterally.
  Interventions: Procedure: GPi-DBS; Device: GPi-DBS devices
- STN-DBS (Experimental): The DBS electrodes are implanted into dorsolateral STN bilaterally.
  Interventions: Procedure: STN-DBS; Device: STN-DBS devices

INTERVENTIONS:
Procedure: GPi-DBS — An elaborate target/trajectory planning and a precise image fusion of MRI and stereotactic CT scanning are performed before surgery. After microelectrode recording, two sets of quadripolar DBS leads (contact interval is 1.5mm) will be inserted into the posteroventral part of bilateral GPi nuclei separately. Subsequently, an implantable pulse generator will be connected via extension wires and implanted at the left/right subclavicular area subcutaneously.
  Arms: GPi-DBS
Procedure: STN-DBS — An elaborate target/trajectory planning and a precise image fusion of MRI and stereotactic CT scanning are performed before surgery. After microelectrode recording, two sets of quadripolar DBS leads (contact interval is 0.5mm) will be inserted into the dorsolateral part of bilateral STN nuclei separately. Subsequently, an implantable pulse generator will be connected via extension wires and implanted at the left/right subclavicular area subcutaneously.
  Arms: STN-DBS
Device: GPi-DBS devices — 1. DBS electrode: 3387 (Medtronic, Minneapolis, MN, USA) or L302 (PINS Medical, Beijing, China) or 1210(SceneRay, Suzhou, China);
  2. Extension wire: 37086 (Medtronic, Minneapolis, MN, USA) or E202 (PINS Medical, Beijing, China) or 1340/SR1341 (SceneRay, Suzhou, China);
  3. Implantable pulse generator: ACTIVA PC/RC (Medtronic, Minneapolis, MN, USA) or G102/G102R (PINS Medical, Beijing, China) or 1180/SR1101 (SceneRay, Suzhou, China).
  Arms: GPi-DBS
Device: STN-DBS devices — 1. DBS electrode: 3389 (Medtronic, Minneapolis, MN, USA) or L301 (PINS Medical, Beijing, China) or 1200 (SceneRay, Suzhou, China);
  2. Extension wire: 37086 (Medtronic, Minneapolis, MN, USA) or E202 (PINS Medical, Beijing, China) or 1340/SR1341 (SceneRay, Suzhou, China);
  3. Implantable pulse generator: ACTIVA PC/RC (Medtronic, Minneapolis, MN, USA) or G102/G102R (PINS Medical, Beijing, China) or 1180/SR1101 (SceneRay, Suzhou, China).
  Arms: STN-DBS

SUMMARY:
Cervical dystonia (CD), also known as spasmodic torticollis, is a type of focal dystonia, mainly manifesting as involuntary head turning or tilting, or holding a twisted posture. Although it can be alleviated by injection of botulinum toxin, the effect is temporary so that patients require multiple injections. Deep Brain Stimulation (DBS) targeting on globus pallidus internus (GPi) or subthalamic nucleus (STN) has been proved to be a safe and effective strategy for primary cervical dystonia, even for those medically refractory cases. However, the question of which target is better has not been clarified.

Therefore, the invstigators design this randomized and controlled trial, aiming to compare the differences between GPi-DBS and STN-DBS for cervical dystonia in the improvement of symptoms , quality of life, mental status, cognitive status, as well as in stimulation parameters and adverse effects. The invstigators hypothesize that STN-DBS will outperform GPi-DBS at short-term follow-up, while the superiority will disappear and the efficacy of the two group will become similar at long-term follow-up.

DETAILED DESCRIPTION:
CD limits the neck activity by involving one or a group of neck muscles and is often accompanied by pain and psychological disorders, seriously affecting the quality of life. GPi and STN are two dominant targets for DBS, either of which has been widely used in the treatment of CD with remarkable efficacy (about 50%-90% symptomatic improvement rate). However, there has been no prospective studies to directly compare the DBS efficacy of these two targets.

The invstigators plan to design a multicenter, prospective, randomized, parallel-controlled equivalent clinical trial, aiming to compare GPi-DBS with STN-DBS for drug-resistant CD in the following aspects: (1) improvement rate of dystonic symptoms, (2) improvement rate of life quality, mental and cognitive status, (3) stimulation parameters, (4) adverse effects.

According to the inclusion and exclusion criteria, a total of 98 idiopathic or hereditary isolated CD patients will be enrolled, each of whom will be randomly divided into GPi-DBS group or STN-DBS group in a 1:1 ratio by central randomization. Informed consent forms are signed and information at baseline is collected. A standardized video will be recorded to assess the severity of the disease. The DBS electrodes will be implanted into posteroventral GPi (GPi-DBS group) or dorsolateral STN (STN-DBS group) respectively. The other operation procedures and subsequent follow-up plan are the same. The DBS device will be switched on in four weeks postoperatively and the optimal stimulation parameters will be used. The invstigators will record standardized videos and/or complete a series of clinical scales (see outcome measures) for all patients at baseline, four weeks postoperatively (after activation of DBS device), three months postoperatively, six months postoperatively, and one year postoperatively. Meanwhile, the stimulation parameters and adverse effects will also be documented. Finally, two professional raters will assess the severity of CD (reflected by Toronto Western Spasmodic Torticollis Rating Scale and Tsui scale) at different timepoints according to those standardized videos in a blind manner.

Intention-to-treatment analysis and per protocol analysis are both conducted by a professional data analyst.

ELIGIBILITY:
Inclusion criteria

1. Diagnosed as idiopathic or hereditary isolated CD;
2. Severe functional impairment;
3. Oral medication and injection of botulinum toxin become ineffective (> 3 months since last injection), or refuse to adopt botulinum toxin injection;
4. No secondary causes of CD;
5. Age 18-80 years old;
6. Normal neurological examination except for dystonia;
7. Normal brain MRI;
8. The subject or their family members can fully understand the trial and sign the informed consent;
9. Good compliance and willingness to receive regular follow-ups.

Exclusion criteria

1. Diagnosed as secondary CD;
2. CD with obvious trunk/limb involvement, or Meige syndrome;
3. History of severe mental disorders, dementia, or epilepsy;
4. Previous dystonia surgery (pallidotomy, thalamotomy, DBS, etc);
5. Accompanied by other neurological diseases (Parkinson's disease, essential tremor, multiple sclerosis, stroke, etc);
6. The patient has or needs other implantable devices (cardiac pacemakers, defibrillators, cochlear implants, spinal cord stimulators, etc);
7. Pregnant women or women who are waiting to become pregnant during the trial;
8. Poor health condition.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Estimated)
Dates: Start 2023-09-01 (Estimated); Primary Completion 2024-12-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Change from baseline Toronto Western Spasmodic Torticollis Rating Scale - Severity subscale (TWSTRS-Severity) at 3 months | Three months postoperatively.
  TWSTRS-Severity subscale can reflect the severity of the dystonia. The total score of TWSTRS-Severity subscale is 35 points. Higher scores indicate more severe symptoms.
Change from baseline Tsui scale at 3 months | Three months postoperatively.
  Tsui scale can better reflect the severity of spasmodic torticollis. It consists of four parts, and the total score was calculated by A*B+C+D. The maximum score was 25 points. After treatment, a 0-10% decrease is considered ineffective, a 11%-50% decrease is considered as partial remission, a 51%-80% decrease is considered as obvious remission, and a 81%-100% decrease is considered as complete remission.
Change from baseline Toronto Western Spasmodic Torticollis Rating Scale - Severity subscale (TWSTRS-Severity) at 6 months | Six months postoperatively.
  TWSTRS-Severity subscale can reflect the severity of the dystonia. The total score of TWSTRS-Severity subscale is 35 points. Higher scores indicate more severe symptoms.
Change from baseline Tsui scale at 6 months | Six months postoperatively.
  Tsui scale can better reflect the severity of spasmodic torticollis. It consists of four parts, and the total score was calculated by A*B+C+D. The maximum score was 25 points. After treatment, a 0-10% decrease is considered ineffective, a 11%-50% decrease is considered as partial remission, a 51%-80% decrease is considered as obvious remission, and a 81%-100% decrease is considered as complete remission.
Change from baseline Toronto Western Spasmodic Torticollis Rating Scale - Severity subscale (TWSTRS-Severity) at 1 year | One year postoperatively.
  TWSTRS-Severity subscale can reflect the severity of the dystonia. The total score of TWSTRS-Severity subscale is 35 points. Higher scores indicate more severe symptoms.
Change from baseline Tsui scale at 1 year | One year postoperatively.
  Tsui scale can better reflect the severity of spasmodic torticollis. It consists of four parts, and the total score was calculated by A*B+C+D. The maximum score was 25 points. After treatment, a 0-10% decrease is considered ineffective, a 11%-50% decrease is considered as partial remission, a 51%-80% decrease is considered as obvious remission, and a 81%-100% decrease is considered as complete remission.

SECONDARY OUTCOMES:
Change of Toronto Western Spasmodic Torticollis Rating Scale - Disability subscale (TWSTRS-Disability) | Three months postoperatively, six months postoperatively, and one year postoperatively.
  TWSTRS-Disability subscale can reflect the disability of the dystonia. The total score of TWSTRS-Disability subscale is 30 points. Higher scores indicate more compromised living ability.
Change of Toronto Western Spasmodic Torticollis Rating Scale - Pain subscale (TWSTRS-Pain) | Three months postoperatively, six months postoperatively, and one year postoperatively.
  TWSTRS-Pain subscale can reflect the level of the neck pain. The total score of TWSTRS-Pain subscale is 20 points. Higher scores indicate more severe neck pain.
Change of 36-item Short Form General Health Survey (SF-36) | Six months postoperatively, and one year postoperatively.
  The SF-36 scale is a comprehensive index that reflects the health status of individuals.This scale has 8 dimensions to evaluate health-related quality of life, namely, physical function (PF), role physical (RP), body pain (BP), general health (GH), vitality (VT), social functioning (SF), role emotional (RE), mental health (MH). Higher score indicates better health status.
Change of Hamilton Anxiety Scale (HAMA) | Six months postoperatively, and one year postoperatively.
  HAMA score can better reflect the severity of anxiety. It is composed of two parts, namely, physical anxiety (item 7-13) and mental anxiety (item 1-6, 14). Total score ≥ 29 points: severe anxiety; Total score ≥21 points: there must be significant anxiety; Total score ≥14 points: there must be anxiety; Total score ≥ 7 points: you may have anxiety; Total score < 7 points: there are no symptoms of anxiety.
Change of 24-item Hamilton Depression Scale (HAMD) | Six months postoperatively, and one year postoperatively.
  HAMD score can better reflect the severity of depression. Total score < 7 points: normal; Total score 7-17 points: possible depression; Total score 17-24 points: definitely depression; Total score > 24 points: severe depression.
Change of Mini-mental State Examination (MMSE) | Six months postoperatively, and one year postoperatively.
  MMSE is a screening scale for Alzheimer's disease. It consists of 20 questions with 30 items (30 points), including five aspects: orientation, memory, attention and calculation, recall, language. Total score > 27 points: normal. Total score 21-27 points: mild cognitive impairment; Total score 10-20 points: moderate cognitive impairment; Total score < 9 points: severe cognitive impairment.
Change of Montreal Cognitive Assessment (MoCA) | Six months postoperatively, and one year postoperatively.
  MoCA is an assessment tool for mild cognitive impairment. The cognitive domains include attention and concentration, executive function, memory, language, visuospatial skills, abstract thinking, calculation and orientation. The total score is 30 points. A score of ≥26 points is considered normal.
Total electrical energy delivered (TEED) | One year postoperatively.
  The formula of TEED is as follows: TEED = Voltage*2*Pulse Width*Frequency/Impedance. The higher the TEED, the shorter the battery life of stimulator.
Adverse effects | Up to 1 year postoperatively.
  Any adverse event occurring between the beginning time of the trial and the last follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Zhiqi Mao, PhD, Principal Investigator — Chinese PLA General Hospital; Bin Liu, MD, Principal Investigator — Chinese PLA General Hospital
Locations (1):
- Chinese PLA General Hospital, Beijing, China

REFERENCES:
- [Derived] Liu B, Xu J, Yang H, Yu X, Mao Z. PAllidal versus SubThalamic deep brain Stimulation for Cervical Dystonia (PASTS-CD): study protocol for a multicentre randomised controlled trial. BMJ Open. 2023 Oct 13;13(10):e073425. doi: 10.1136/bmjopen-2023-073425. PMID 37832982